CLINICAL TRIAL: NCT00098033
Title: Phase II Clinical and Pharmacodynamic Investigation of Clofarabine in Acute Leukemias
Brief Title: Investigation of Clofarabine in Acute Leukemias
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas (Other)
Organization: FDA Office of Orphan Products Development (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2127
Record Dates: First submitted 2004-12-02; First posted 2004-12-03 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2004-12

CONDITIONS: Acute Myelogenous Leukemia; Acute Lymphocytic Leukemia; Chronic Myelogenous Leukemia
Keywords: clinical; pharmacodynamics; investigational drug clofarabine; AML, ALL, CML-accelerated phase, CML-blastic phase; Chronic Myelogenous Leukemia - accelerated phase; Chronic Myelogenous Leukemia - blastic phase
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myeloid, Accelerated Phase; Blast Crisis | interventions — Clofarabine

INTERVENTIONS:
Drug: clofarabine

SUMMARY:
The goals and objectives of this project are to evaluate the antileukemic activity of the investigational agent clofarabine in patients with acute myelogenous leukemia (AML), acute lymphocytic leukemia (ALL), and chronic myelogenous leukemia (CML) in accelerated and blastic phases.

DETAILED DESCRIPTION:
The specific aims of the project are (1) conduct the phase II study of clofarabine and evaluate the antileukemic efficacy in AML, ALL, and CML-accelerated and blastic phases in terms of complete response (CR) rate, response duration, and survival; and (2) analyze the relationship between cellular uptake and retention of clofarabine triphosphate (the active metabolite), inhibition of DNA synthesis, and clinical outcome.

Completion date provided represents the completion date of the grant per OOPD records

ELIGIBILITY:
* Patient is diagnosed with AML, ALL, myelodysplastic syndrome (MDS), and CML in transformation (includes CML-blastic phase and CML-accelerated phase).
* No prior chemo-, immuno-, or radio-therapy for 2 weeks before entering the study, unless progressive life-threatening leukemia as judged by the treated physician.
* Adequate liver function (bilirubin </= 2 mg%) and renal function (creatinine </= 2 mg%).
* Pregnant and lactating females not eligible.
* Zubrod performance status 0-2
* Adequate cardiac status
* No life-threatening conditions (e.g. infections) which may cause death within 3 weeks.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 64
Dates: Start 2002-09; Study Completion 2005-09

CONTACTS AND LOCATIONS:
Overall Officials: Hagop M Kantarjian, MD, Principal Investigator — M.D. Anderson Cancer Center; Jorge E Cortes, MD, Study Chair — M.D. Anderson Cancer Center

REFERENCES:
- [Background] Cortes JE, Gandhi V, et al. Clofarabine (2-chloro-9-(deoxy-2-fluoro-b-D-arabinosfuranosyl)adenine) is active for patients with refractory or relapsed acute leukemia. #739 ASH 2002.
- See also: FDA's clinical trials website — http://www.clinicaltrials.gov